CLINICAL TRIAL: NCT06229834
Title: Chiropractic Care for Episodic Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Palmer College of Chiropractic (Other); Yale University (Other); VA Connecticut Healthcare System (U.S. Federal Agency); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Peter M. Wayne, Ph.D., Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023P003554; R01AT012228-01 (NIH)
Record Dates: First submitted 2024-01-12; First posted 2024-01-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Episodic Migraine
Keywords: migraine; headache disorder
MeSH Terms: conditions — Migraine Disorders; Headache Disorders

STUDY DESIGN:
Intervention Model Description: A two-arm pilot randomized attention-controlled trial at two sites which are representative of sites to be included in the future large-scale trial (Osher Clinic, BWH, and VA Medical Center, West Haven, CT). We will recruit and randomize 60 individuals (30 per site). Individuals will be randomized (1:1) to: 1) 14 sessions of CC (6 sessions of chiropractic care over 3-5 weeks followed by 8 sessions of chiropractic care (CC) over 12 weeks); or 2) 14 sessions of headache health education (15-minute 1:1 virtual sessions focused on pre-defined migraine-specific topics) - both added to usual medical care. Individuals will be followed for 4 weeks after the end of their intervention period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: While participants, treating chiropractors, study coordinators, and research assistants will be unblinded to treatment assignment, study investigators who are not involved in providing chiropractic care treatments or monitoring adverse events will be blinded. The blinding of these investigators and the programmer will only be broken after approval of the final statistical analysis plan and locking of the trial data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiropractic Care (Experimental): 4 sessions of chiropractic care (6 sessions of chiropractic care over 3-5 weeks followed by 8 sessions of chiropractic care over 12 weeks); participants will be allowed to continue usual care throughout the study.
  Interventions: Procedure: Chiropractic Care
- Headache Health Education (HHE) (Other): Participants randomized to Headache Health Education (HHE) will receive 14 interactive 15-minute education sessions delivered via videoconference.
  Interventions: Behavioral: Headache Health Education

INTERVENTIONS:
Procedure: Chiropractic Care — The chiropractic care protocol can be personalized to the patient's clinical needs and follows the scope of chiropractic care practice in the Commonwealth of Massachusetts and the State of Connecticut. Components of the chiropractic intervention include: posture correction / spinal stabilization exercises; soft tissue relaxation techniques; spinal manipulation (i.e. chiropractic adjustment) / mobilization; breathing and relaxation techniques; stretches, self-care; ergonomic modifications; bracing and supports.
  Arms: Chiropractic Care
Behavioral: Headache Health Education — Participants randomized to the HHE arm will receive 14 interactive 15-minute education sessions delivered via video conference.
  To partially control for attention and expectation associated with chiropractic care, participants randomized to the control group will receive a modified version of a headache education intervention we employed in our pilot study. Participants randomized to HHE will receive 14 interactive 15-minute education sessions delivered via VA or MGB Teams. Material to be covered will focus on pre-defined migraine-specific topics, compared with the control for our pilot study, in addition to greater contact time, HHE will be delivered in a more interactive manner utilizing active learning principles known to support adult learning. We will also utilize publicly available short videos (e.g., from the American Headache Society) followed by scripted discussions with the participant. Example topics include the physiology of migraine or the contribution of life.
  Arms: Headache Health Education (HHE)

SUMMARY:
Migraine, a chronic intermittent headache disorder, ranks in the top five causes of years lived with disability. One promising non-pharmacologic and integrative treatment for migraine may be chiropractic care due to the co-occurrence of migraine and musculoskeletal complaints. The goal of this application is to perform a pilot study of chiropractic care for episodic migraine to help inform the design of a future, full-scale pragmatic effectiveness trial.

DETAILED DESCRIPTION:
Migraine, a chronic intermittent headache disorder, ranks in the top five causes for years lived with disability. Due to the high disability burden associated with migraine, individuals who experience migraine often seek treatments to reduce the frequency and severity of their attacks and often express interest in nonpharmacologic and integrative approaches. One promising treatment may be chiropractic care due to the comorbidity of migraine and musculoskeletal complaints.

Our long-term goal is to conduct a multi-site large-scale, fully powered trial evaluating the effectiveness of a validated multimodal chiropractic care intervention to reduce migraine frequency, severity, and disability.

To help inform the design of a large-scale trial with both pragmatic and explanatory features, we propose to conduct a two-arm pilot randomized attention-controlled trial at two sites which are representative of sites to be included in the future large-scale trial. We will recruit and randomize 60 individuals (30 per site) to either 1) 14 visits of chiropractic care (CC) (6 visits of CC over 3-5 weeks followed by 8 visits of CC over 12 weeks); or 2) 14 sessions of headache health education (15-minute 1:1 virtual sessions focused on pre-defined migraine specific topics) - both added to usual medical care. This study will allow us to address the following aims: 1) To train a team of chiropractors from established clinics within two academic medical centers with existing partnerships with headache programs, refine our intervention, and assess the fidelity of intervention protocols; 2) To optimize data collection, data management, and reporting procedures across sites and establish the infrastructure needed for a large-scale trial; 3) To assess the feasibility of recruitment, retention, and adherence across multiple study sites; 4) To assess participant expectations and treatment experience.

ELIGIBILITY:
Inclusion Criteria

* Age 18-65 years
* Confirmed diagnosis of migraine with or without aura which does not meet criteria for chronic migraine according to the International Classification for -Headache Disorders (ICHD)-3 guidelines at the screening visit with the study physician
* History of migraines dating for at least one year
* Completion of at least 26 headache diary days out of 28
* Confirmed migraine frequency ≥4 to ≤13 days per month during a run-in period
* If use of medication is applicable, dose must be stable for 2 months prior to study enrollment
* If use of medication for non-migraine pain condition is applicable (with the exception of episodic tension type headache), dose must be stable for 2 months prior to study enrollment
* Willing and able to complete all study procedures and be randomized to either of the two intervention groups
* Fluency in English
* Confirmed access to and proficiency with use of a smartphone, computer, and/or tablet
* Working email address or willingness to create an email account for the study

Exclusion Criteria

* Non-Veterans (VAMC only)
* Received botulinum toxin treatment for headache and/or neck pain within the 4 months prior to the start of the baseline phase
* Received chiropractic care for any condition within the 3 months prior to the start of the baseline phase
* Received behavioral interventions (e.g., cognitive behavioral therapy, acceptance and commitment therapy, mindfulness, relaxation techniques, hypnosis) within the past 3 months)
* Used neuromodulation (i.e., "headache devices"), procedures for migraine prevention within the 2 months before the baseline period, or investigational medications or headache devices for at least 90 days prior to screening
* Diagnosis of medication overuse headache according to the ICHD-3 guidelines at the screening visit with the study physician
* Traumatic Brain Injury ≤ 1 year before screening visit or worsening of migraine as noted by the screening study physician
* Head or neck trauma within the past year causing neurological or musculoskeletal signs or symptoms requiring treatment
* Any medical, neurologic, or psychiatric condition that the screening study physician deems would lead to difficulty complying with the protocol or negatively impact the safety profile of the interventions
* Psychiatric hospitalization in the last 6 months
* Receiving hospice or palliative care
* History of carotid or vertebral artery dissection
* Presence of carotid bruits
* Presence of contraindications (relative or absolute) for spinal manipulation or mobilization where these procedures cannot be modified for safe administration and are consistent with those published by the World Health Organization (WHO) guidelines, including but not limited to:
* Local spinal hypermobility/instability
* Conditions causing general spinal hypermobility, such as Marfan, Ehlers-Danlos syndrome, and Osteogenesis imperfecta
* Malignancy of the spine or spinal cord
* Frank disc herniation with signs of progressive neurological deficit
* Spinal or intracanalicular hematomas Inflammatory spondyloarthropathies such as rheumatoid arthritis
* Spinal fractures or dislocations
* Avascular necrosis in an area of proposed joint manipulation
* Bone-weakening disorders affecting the spine, such as benign bone tumors, infection, or osteoporosis
* Vertebrobasilar insufficiency syndrome
* Aneurysm involving a major blood vessel in an area of potential joint manipulation
* History of stroke
* Anticoagulant therapy or blood disorders cause significant bleeding tendency
* Cervical spine congenital anomalies that affect the stability or neurologic integrity of the individual or history of cervical spine surgery
* Either self-reported current alcohol or substance use disorder or current alcohol or substance use disorder documented by a treating medical provider within the past 6 months
* Hormone replacement therapy for less than six months, or if prescriptions greater than 6 months in duration must be at a stable dose
* Significant cognitive impairment that would impair participation in the trial
* Currently pregnant or intention to become pregnant within the next six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility (average number of participants per month) | 16 months
  Each site will be able to recruit 30 participants within 16 months
Retention feasibility (proportion of participants not lost to follow-up) | 20 weeks
  Retention will be quantified by the proportion of subjects who record their migraines for at least 26 out of 28 days and all questionnaires at each outcome assessment.
Intervention adherence feasibility | 15 weeks
  Adherence will be calculated as the proportion of subjects who attend at least 80% of the chiropractic care visits or 80% of the one-on-one headache health education video-conferences.

SECONDARY OUTCOMES:
Number of days with migraine headaches | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  Number of migraine headaches as recorded in migraine diaries.
Proportion of responders | Change from baseline to initial follow-up (16 weeks) and change from baseline to final follow-up (20 weeks).
  Proportion of individuals who experience a ≥50% reduction in migraine days.
Average severity of migraine attacks | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  Average severity of migraine attacks (on a 1 to 10 scale) as recorded in migraine diaries.
Average number of hours for a migraine attack (duration) | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  Average number of hours a migraine attack lasted as recorded in migraine diaries.
Average number of medications used for a migraine attack | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  Average number of medications used to treat a migraine attack as recorded in migraine diaries
Neck Disability Index (NDI) | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  Self-report questionnaire used to determine how neck pain impacts daily activities of living and self-related neck pain disability.
  Score range: 10 - 60. Higher scores indicate greater disability.
Headache Related Disability (HIT-6) | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  HIT-6 is a validated 6-item assessment that evaluates the impact headaches have on a participant's life. Score range: 36 - 78. Higher scores indicate greater disability.
Migraine Specific Quality of Life Questionnaire, version 2.1 (MSQv2.1) | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  Migraine Specific Quality of Life Questionnaire, version 2.1 (MSQv2.1) is a validated 14-item questionnaire; it is one of the most frequently used disability instrument in migraine research and is highly reliable.
  Participants are asked to provide their response to each question using a standard six point Likert-type scale (none of the time; a little bit of the time; some of the time; a good bit of the time; most of the time; all of the time). Each MSQoL v.2.1 dimension is scored independently from 0 to 100 such that a higher score indicates a better quality of life.
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  PROMIS-29 is a system of validated, highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being.
  PROMIS-29 v2. 0 profile measure assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items for each domain.The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
PTSD Checklist for DSM-5 (PCL-5) | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  20-item self-report measure of the DSM-5 symptoms of PTSD. Score range: 0 - 5. Higher scores are associated with greater likelihood of PTSD.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Assess during three 4-week periods (baseline, initial follow-up, final follow-up) within the total of 24 weeks that participants are enrolled in the trial.
  Godin Leisure-Time Exercise Questionnaire will be used to measure the amount and intensity of general exercise during the study period. This validated instrument consists of 4 items measuring the frequency of light, moderate, and vigorous-intensity leisure-time physical activity. In the GLTEQ, individuals are asked to complete a self-explanatory, brief four-item query of usual leisure-time exercise habits.
  Higher score indicate more leisure-time exercise per week.
The Expectations for Complementary and Alternative Medicine Treatments Questionnaire short form (EXPECT) | Assess only at baseline following the 4 weeks run-in phase but before randomization.
  EXPECT Questionnaire (short form) is a recently developed and validated questionnaire used to assess individuals' expectations of treatments for chronic pain.
  Score range: 0 - 40. Higher scores indicate higher expectation of recovery after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Osher Center for Integrative Health, Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Investigators interested in using data from this trial will be directed to contact the multiple principle investigators for data access.

REFERENCES:
- [Background] Albrecht DS, Mainero C, Ichijo E, Ward N, Granziera C, Zurcher NR, Akeju O, Bonnier G, Price J, Hooker JM, Napadow V, Loggia ML, Hadjikhani N. Imaging of neuroinflammation in migraine with aura: A [11C]PBR28 PET/MRI study. Neurology. 2019 Apr 23;92(17):e2038-e2050. doi: 10.1212/WNL.0000000000007371. Epub 2019 Mar 27. PMID 30918090
- [Background] Arnold M, Kappeler L, Georgiadis D, Berthet K, Keserue B, Bousser MG, Baumgartner RW. Gender differences in spontaneous cervical artery dissection. Neurology. 2006 Sep 26;67(6):1050-2. doi: 10.1212/01.wnl.0000237341.30854.6a. PMID 17000975
- [Background] Ashina S, Bendtsen L, Lyngberg AC, Lipton RB, Hajiyeva N, Jensen R. Prevalence of neck pain in migraine and tension-type headache: a population study. Cephalalgia. 2015 Mar;35(3):211-9. doi: 10.1177/0333102414535110. Epub 2014 May 22. PMID 24853166
- [Background] Beaton-Starr M, Rist PM, Connor JP, Wayne PM, Osypiuk K, Bernstein C. Development and Implementation of the Integrative Toolbox for Headache Management. Headache. 2020 Apr;60(4):771-775. doi: 10.1111/head.13743. Epub 2020 Jan 9. PMID 31919834
- [Background] Befus DR, Hull S, Strand de Oliveira J, Schmidler GS, Weinberger M, Coeytaux RR. Nonpharmacological Self-Management of Migraine Across Social Locations: An Equity-Oriented, Qualitative Analysis. Glob Adv Health Med. 2019 Jun 13;8:2164956119858034. doi: 10.1177/2164956119858034. eCollection 2019. PMID 31223518
- [Background] Bernstein C, Wayne PM, Rist PM, Osypiuk K, Hernandez A, Kowalski M. Integrating Chiropractic Care Into the Treatment of Migraine Headaches in a Tertiary Care Hospital: A Case Series. Glob Adv Health Med. 2019 Mar 28;8:2164956119835778. doi: 10.1177/2164956119835778. eCollection 2019. PMID 30944771
- [Background] Connor JP, Bernstein C, Kilgore K, Rist PM, Osypiuk K, Kowalski M, Wayne PM. Perceptions of Chiropractic Care Among Women With Migraine: A Qualitative Substudy Using a Grounded-Theory Framework. J Manipulative Physiol Ther. 2021 Feb;44(2):154-163. doi: 10.1016/j.jmpt.2020.07.001. Epub 2021 Jan 9. PMID 33431279
- [Background] Lisi AJ, Brandt CA. Trends in the Use and Characteristics of Chiropractic Services in the Department of Veterans Affairs. J Manipulative Physiol Ther. 2016 Jun;39(5):381-386. doi: 10.1016/j.jmpt.2016.04.005. PMID 27288324
- [Background] Rist PM, Bernstein C, Kowalski M, Osypiuk K, Connor JP, Vining R, Long CR, Macklin EA, Wayne PM. Multimodal chiropractic care for migraine: A pilot randomized controlled trial. Cephalalgia. 2021 Mar;41(3):318-328. doi: 10.1177/0333102420963844. Epub 2020 Oct 13. PMID 33050719
- [Background] Rist PM, Buring JE, Ridker PM, Kase CS, Kurth T, Rexrode KM. Lipid levels and the risk of hemorrhagic stroke among women. Neurology. 2019 May 7;92(19):e2286-e2294. doi: 10.1212/WNL.0000000000007454. Epub 2019 Apr 10. PMID 30971484
- [Background] Rist PM, Hernandez A, Bernstein C, Kowalski M, Osypiuk K, Vining R, Long CR, Goertz C, Song R, Wayne PM. The Impact of Spinal Manipulation on Migraine Pain and Disability: A Systematic Review and Meta-Analysis. Headache. 2019 Apr;59(4):532-542. doi: 10.1111/head.13501. Epub 2019 Mar 14. PMID 30973196
- [Background] Wayne PM, Bernstein C, Kowalski M, Connor JP, Osypiuk K, Long CR, Vining R, Macklin E, Rist PM. The Integrative Migraine Pain Alleviation through Chiropractic Therapy (IMPACT) trial: Study rationale, design and intervention validation. Contemp Clin Trials Commun. 2020 Jan 22;17:100531. doi: 10.1016/j.conctc.2020.100531. eCollection 2020 Mar. PMID 32043014
- [Background] Wayne PM, Buring JE, Davis RB, Connors EM, Bonato P, Patritti B, Fischer M, Yeh GY, Cohen CJ, Carroll D, Kiel DP. Tai Chi for osteopenic women: design and rationale of a pragmatic randomized controlled trial. BMC Musculoskelet Disord. 2010 Mar 1;11:40. doi: 10.1186/1471-2474-11-40. PMID 20193083
- [Background] Wayne PM, Gagnon MM, Macklin EA, Travison TG, Manor B, Lachman M, Thomas CP, Lipsitz LA. The Mind Body-Wellness in Supportive Housing (Mi-WiSH) study: Design and rationale of a cluster randomized controlled trial of Tai Chi in senior housing. Contemp Clin Trials. 2017 Sep;60:96-104. doi: 10.1016/j.cct.2017.07.005. Epub 2017 Jul 8. PMID 28694204
- [Background] Wayne PM, Manor B, Novak V, Costa MD, Hausdorff JM, Goldberger AL, Ahn AC, Yeh GY, Peng CK, Lough M, Davis RB, Quilty MT, Lipsitz LA. A systems biology approach to studying Tai Chi, physiological complexity and healthy aging: design and rationale of a pragmatic randomized controlled trial. Contemp Clin Trials. 2013 Jan;34(1):21-34. doi: 10.1016/j.cct.2012.09.006. Epub 2012 Sep 29. PMID 23026349